CLINICAL TRIAL: NCT05142683
Title: Effectiveness of an Integrated Care Pathway for Adolescent Depression: A Quasi-experimental, Multi-site, Cluster Controlled Trial (Edited on March 7th, 2024)
Brief Title: Effectiveness of an Integrated Care Pathway for Depression: Cluster Randomized Controlled Trial
Acronym: CARIBOU-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); The Hospital for Sick Children (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 019/2021
Record Dates: First submitted 2021-11-03; First posted 2021-12-02 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Major Depressive Disorder
Keywords: Adolescents; Integrated Care Pathway; Depression; Measurement Based Care; Implementation
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: The study uses a Type 1 Hybrid Implementation Effectiveness design that focuses on the effectiveness of the clinical intervention (ICP) while exploring the implementation effectiveness of the intervention.
  A stepped wedge, cluster randomized controlled trial is indicated as the intervention is applied at the clinic level.
  Edited on March 7th, 2024: The study uses a Type 1 Hybrid Implementation Effectiveness design that focuses on the effectiveness of the clinical intervention (ICP) while exploring the implementation effectiveness of the intervention.
  A cluster controlled trial is indicated as the intervention is applied at the clinic-level.
Who Masked: Outcomes Assessor
Masking Description: The evaluator of the primary outcome will be blind to treatment arm as well as blind to the stepped wedge design.
  Edited March 7th, 2024: The evaluator of the primary outcome will be blind to treatment arm as well as blind to the quasi-experimental cluster controlled design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (Active Comparator): Study involvement for all sites will begin in the TAU condition, which is the typical treatment at the participating community mental health agency. A range of treatments observed in our previous survey of sites will be on offer in these agencies, depending on the preferences and context of the local agency. In typical TAU in community mental health agencies, depressive symptoms and function are not systematically monitored via standardized rating scales. TAU may or may not include referral to psychotherapy and/or parent support. There are no prompts to prescribe specific medications, and/or internal and external referrals to treatment and other services, guided by local service standards.
  Interventions: Other: Treatment As Usual
- CARIBOU-2 (Experimental): After the CARIBOU-1 pilot study, the Principal Investigator revised the ICP to render it more applicable to community settings as well as offer a second-line psychotherapy ("Brief Psychosocial Intervention") for youth who do not engage with, or respond to, cognitive-behavioural therapy. The revised version is called the CARIBOU-2 intervention. The current iteration of the pathway involves a series of steps: (1) structured assessment, including safety assessment; (2) education on depression, sleep, exercise, and diet; (3) psychotherapy (with 1st line Cognitive Behavioural Therapy, 2nd line "Brief Psychosocial Intervention"); (4) a caregiver structured support group; (5) medication options (1st line fluoxetine, 2nd line sertraline); (6) "team reviews" every four weeks, (meeting with the youth and involved clinicians to review measures and discuss treatment changes); and, (7) discharge and follow-up planning.
  Interventions: Other: CARIBOU-2

INTERVENTIONS:
Other: Treatment As Usual — Various typical interventions for adolescents with depression.
  Arms: Treatment as Usual
Other: CARIBOU-2 — Integrated Care Pathway intervention for adolescents with depression.
  Arms: CARIBOU-2

SUMMARY:
This a stepped wedged cluster RCT with two intervention arms--Treatment As Usual (TAU) and an Integrated Care Pathway (ICP). Eligible participants are between the ages of 13 and 18, who present to community mental health agencies with depressive symptoms as the primary concern. The primary objective is to establish the clinical effectiveness of the ICP intervention in the community setting relative to TAU, with respect to reducing evaluator-rated depressive symptoms. The secondary objectives are to explore changes in clinician-rated function and caregiver-rated symptoms for youth receiving the ICP intervention relative to TAU. The third objective is to explore the implementation effectiveness of the ICP intervention, namely investigating: feasibility, fidelity, cost and acceptability.

Edited on March 7th, 2024: This is a quasi-experimental, multi-site cluster controlled clinical trial design with two intervention arms--Treatment As Usual (TAU) and an Integrated Care Pathway (ICP). Eligible participants are between the ages of 13 and 18, who present to community mental health agencies with depressive symptoms as the primary concern. The primary objective is to establish the clinical effectiveness of the ICP intervention in the community setting relative to TAU, with respect to reducing evaluator-rated depressive symptoms. The secondary objectives are to explore changes in clinician-rated function and caregiver-rated symptoms for youth receiving the ICP intervention relative to TAU. The third objective is to explore the implementation effectiveness of the ICP intervention in the community setting, namely investigating: feasibility, fidelity, cost and acceptability.

DETAILED DESCRIPTION:
Background: Depression is the leading cause of disability in adolescents and a potent risk factor for adolescent suicide. Evidence-based treatments are available; however, many clinics do not provide guidelines-based treatments. Integrated Care Pathways (ICPs) are treatment algorithms based on the highest quality practice guidelines intended to facilitate the delivery of evidence-based treatment at the clinic level. Our group has already tested the feasibility of ICP for adolescent depression at an academic setting. There is still uncertainty regarding whether ICPs lead to improved outcomes in adolescent depression in community setting relative to typical care.

Objective: The current study aim is to test the effectiveness of an ICP for depression in adolescents, called the CARIBOU-2 intervention, versus treatment-as-usual (TAU) in community settings. We hypothesize that participants receiving the ICP will show greater clinical improvement (in symptoms and functioning) than participants in TAU. This study will also examine important implementation outcomes.

Method: The primary participants will be adolescents (N= 648), between the ages of 13 to 18 with depressive symptoms, presenting to one of six selected community mental health agencies. Through a stepped wedge design, all sites will begin in the TAU condition and transition to the ICP condition in a randomized sequence. The primary clinical outcome of interest is the difference between treatment groups in the rate of change of depressive symptoms from baseline to 24-week endpoint as measured by the Childhood Depression Rating Scale-Revised. Secondary outcomes include rate of change of functional improvement, as measured by the Children's Global Assessment Scale, and caregiver-rated internalizing symptoms as rated by the Childhood Behaviour Checklist.

Generalized linear mixed-effects model is a proper choice to test our clinical hypotheses to control for covariates (e.g. demographics and baseline clinical measures), to accommodate multiple forms of the outcome (e.g. continuous, categorical and count type), and to account for clustering at individual level (for repeated measures) and at site level. Time, stage assignment and their interactions will serve as the primary predictors for the analyses. As an example, if we let Y_ijt to denote a continuous outcome of the j-th participant of the i-th site measured at time t, a linear model for Y_ijt will look like the following:

Y_ijt=β_0+〖b_(0,ij)+b_(1,i)+β〗_1 t+β_2 〖Group〗_(i,t)+β_3 Group_it*t+〖β_4 X_ijt+ϵ〗_ijt

of which 〖Group〗_(i,t) denotes the treatment assignment of the i-th site at time t, X_ijt, additional covariates, b_(0,ij) and b_(1,i), random effects at individual and site levels respectively, ϵ_( ijt), unexplained random error, and β's, regression coefficients. For sensitivity analyses, we will explore the use of quadratic or piecewise models when the linear model may not be adequate. We will adopt the intention-to-treat approach in general and use multiple imputation methods as the primary missing data strategy.

Count data, proportions and qualitative data will be used to describe implementation outcomes.

Relevance: Should our results be consistent with our hypotheses, systematic implementation of the CARIBOU-2 intervention to other community mental health agencies would be indicated.

Edited on March 7th, 2024

Background: Depression is the leading cause of disability in adolescents and a potent risk factor for suicide. Evidence-based treatments are available; however, many clinics do not provide guidelines-based treatments. Integrated Care Pathways (ICPs) are treatment algorithms based on the highest quality practice guidelines intended to facilitate the delivery of evidence-based treatment at the clinic level. Our group has already tested the feasibility of ICP for adolescent depression at an academic setting. There is still uncertainty regarding whether ICPs lead to improved outcomes in depression in adolescents in community settings relative to typical care.

Objective: The current study aim is to test the effectiveness of an ICP for depression in adolescence, called the CARIBOU-2 intervention, versus treatment-as-usual (TAU) in community settings. This study will also examine important implementation outcomes.

Method: The primary participants will be adolescents (N= 300 ), between the ages of 13 to 18 with depressive symptoms, presenting to one of six selected community mental health agencies. Through a quasi-experimental, multi-site cluster controlled clinical trial design, sites will begin in the TAU condition and transition to the ICP condition once local enrollment to TAU has reached 25 participants. . The primary clinical outcome of interest is the difference between treatment groups in the rate of change of depressive symptoms from baseline to 24-week endpoint as measured by the Childhood Depression Rating Scale-Revised. Secondary outcomes include rate of change of functional improvement, as measured by the Children's Global Assessment Scale, and caregiver-rated internalizing symptoms as rated by the Childhood Behaviour Checklist. This study will also be examining the following implementation outcomes: feasibility, fidelity cost and acceptability.

Generalized linear mixed-effects model will be the primary analytic tool for evaluating whether the CARIBOU-2 intervention is more effective than TAU for adolescents with depression presenting to care in the community with regards to improvement of depressive symptoms (Hypothesis A), self-reported functioning (Hypothesis B), caregiver-reported internalizing psychopathology (Hypothesis C), and suicidal ideation and behaviours (exploratory). Generalized linear mixed-effects model is a proper choice to control for covariates (e.g. demographics and baseline clinical measures), to accommodate multiple forms of the outcome (e.g. continuous, categorical and count type), and to account for clustering at individual level (for repeated measures) and at site level. Time, treatment assignment and their interactions will serve as the primary predictors for the analyses. As an example, if we let Y_ijt to denote a continuous outcome of the j-th participant of the i-th site measured at time t, a linear model for Y_ijt will look like the following:

Y_ijt=β_0+〖b_(0,ij)+b_(1,i)+β〗_1 t+β_2 〖Group〗_(i,t)+β_3 Group_it*t+〖β_4 X_ijt+ϵ〗_ijt

of which 〖Group〗_(i,t) denotes the treatment assignment of the i-th site at time t, X_ijt, additional covariates, b_(0,ij) and b_(1,i), random effects at individual and site levels respectively, ϵ_( ijt), unexplained random error, and β's, regression coefficients. For sensitivity analyses, we will explore the use of the piecewise model to model the time trend differently . We will adopt the intention-to-treat approach in general and use multiple imputation methods as the primary missing data strategy.

Count data, proportions and qualitative data will be used to describe implementation outcomes.

Relevance: Should our results be consistent with our hypotheses, systematic implementation of the CARIBOU-2 intervention to other community mental health agencies would be indicated.

ELIGIBILITY:
Inclusion Criteria:

* Youth is aged 13 to 18 years, inclusive.
* Youth and/or their caregiver is expressing that 'depression" (or some synonym) is a concern.
* Clinician agrees that depressive symptoms are a treatment target.
* Mood and Feelings Questionnaire score is ≥22 at two sequential visits (screening and baseline assessment).
* Youth must be new to the site (in past 3 months) or have a period of no treatment for 3 months

Exclusion Criteria:

* Known or highly suspected presentations of psychotic symptoms that are persistent, affect functioning, and have observable effects on behaviour.
* Severe substance use disorder, bipolar disorder, autism spectrum disorder or intellectual disability, severe eating disorder, imminent risk of suicide requiring hospitalization as per judgment of the assessing clinician.
* Inability to provide informed consent to the study for any reason
* Youth currently in Day Treatment

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Childhood Depression Rating Scale-Revised | Change from baseline to 24 weeks
  A 17-item measure rated by an RA following a semi-structured interview with the adolescent relating to symptoms of depression over the past 2 weeks. The RA will be blind to treatment assignment.

SECONDARY OUTCOMES:
Columbia Suicide Severity Rating Scale | Change from baseline to 24 weeks
  This measure contains items related self-injurious thoughts and behaviours. RAs rate 3 subscales: Suicidal Ideation Severity, Suicidal Behaviour (which includes suicide attempts and an item for non-suicidal self-injury that is recorded as distinct from suicidal behaviour), and Lethality.
Depression Rating Scale | Change from baseline to 24 weeks
  This is an RA-rated 13-item subscale found in the Kiddie Schedule for Affective Disorders and Schizophrenia-Lifetime version used to assess for DSM-5 criteria of Major Depressive Disorder.
Youth Quality of Life Scale Research Version | Change from baseline to 24 weeks
  This is a 41 item self-report scale measuring the broad array of constructs including sense of self-worth, quality of relationships, sense of agency and life satisfaction.
Health and Social Service Utilization | Change from baseline to 24 weeks
  This is a 10-item, self-report questionnaire that collects data regarding services and medications used by the patient.
Ontario Perception of Care Tool for Mental Health and Addictions | Change from baseline to 24 weeks
  Two versions of this tool were developed by CAMH (one for registered patients and one for family members of clients) and typically consists of 38 items on a Likert scale. It standardizes how substance use, mental health, and concurrent disorder services obtain client perception of care feedback.
Adolescent Alcohol and Drug Involvement Scale Grid | Change from baseline to 24 weeks
  This scale is used for adolescent substance abuse frequency. It includes both alcohol and other drug abuse.
Cognitive Behavioural Therapy Skills Questionnaire | Change from baseline to 24 weeks
  This 16-item measure utilizing a Likert scale from 1 (I don't do this) to 5 (I always do this) assess an individual's cognitive restructuring and behavioral activation skills.
CollaboRATE | Change from baseline to 24 weeks
  This is a 3 item measure on a 5-point Likert Scale that measures the level of shared decision making in the clinical encounter from the patient's perspective, as part of assessing health care quality and provider performance.
Nonsuicidal Self-Injury | Change from baseline to 24 weeks
  This measure comes from the Self-Injurious Thoughts and Behaviors Interview, which is a structured interview that assesses the presence, frequency, and characteristics of a wide range of self-injurious thoughts and behaviors, including suicidal ideation, suicide plans, suicide gestures, suicide attempts, and nonsuicidal self-injury (NSSI). The NSSI section has been adapted for the purposes of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Darren B Courtney, MD, Principal Investigator — University of Toronto
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bennett K, Courtney D, Duda S, Henderson J, Szatmari P. An appraisal of the trustworthiness of practice guidelines for depression and anxiety in children and youth. Depress Anxiety. 2018 Jun;35(6):530-540. doi: 10.1002/da.22752. Epub 2018 Apr 26. PMID 29697887
- [Background] Courtney D, Bennett K, Henderson J, Darnay K, Battaglia M, Strauss J, Watson P, Szatmari P. A Way through the woods: Development of an integrated care pathway for adolescents with depression. Early Interv Psychiatry. 2020 Aug;14(4):486-494. doi: 10.1111/eip.12918. Epub 2019 Dec 27. PMID 31883210
- [Background] Courtney DB, Bennett K, Szatmari P. The Forest and the Trees: Evidence-Based Medicine in the Age of Information. J Am Acad Child Adolesc Psychiatry. 2019 Jan;58(1):8-15. doi: 10.1016/j.jaac.2018.06.035. PMID 30577942
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Derived] Hytman L, Mansueto S, Chan JI, Kumar R, Nguyen ATP, Wang W, Krause KR, Monga S, Szatmari P, Courtney DB. Interrater Reliability and Measurement Error of the Children's Depression Rating Scale-Revised in Adolescents. JAACAP Open. 2025 Jun 20;3(4):1225-1235. doi: 10.1016/j.jaacop.2025.06.005. eCollection 2025 Dec. PMID 41367969
- [Derived] de Oliveira C, Mason J, Amani B, Liddell G, Szatmari P, Henderson J, Courtney D. Protocol for the economic evaluation of the Care for Adolescents who Received Information 'Bout Outcomes, 2nd iteration (CARIBOU-2) non-randomised, cluster-controlled trial of an integrated care pathway for depression in adolescents. BMJ Open. 2025 May 15;15(5):e092541. doi: 10.1136/bmjopen-2024-092541. PMID 40379352